CLINICAL TRIAL: NCT02410980
Title: In-vivo Non-invasive Skin Imaging Pilot Study to Assess the Effects of Tretinoin Cream Using Multi-photon Microscopy and Multi-spectral Imaging
Brief Title: Assessing the Effects of Tretinoin Cream on Human Skin With Optical Imaging Technologies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Unilever R&D (Industry); Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Mihaela Balu, Ph.D. Associate Specialist, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20141508
Record Dates: First submitted 2015-03-23; First posted 2015-04-08 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Collagen Fibril Alteration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tretinoin cream 0.1% (Experimental): Assessment of the skin change
  Interventions: Drug: Tretinoin cream 0.1%

INTERVENTIONS:
Drug: Tretinoin cream 0.1% — Assessment of the skin change

SUMMARY:
The researchers will assess the effects of treatment with tretinoin cream on human skin by using non-invasive optical imaging technologies.

DETAILED DESCRIPTION:
The researchers will evaluate changes in the dermis and skin properties as the effect of treatment with Tretinoin cream (0.1%) by using the following optical imaging techniques.

1. Multiphoton microscopy using a clinical tomograph (MPTflex, Jenlab, Germany)
2. Multispectral Imaging using a device developed at Beckman Laser Institute, UC Irvine

ELIGIBILITY:
Inclusion Criteria:

* Female 45 years of age or older - Skin type scale I to III

Exclusion Criteria:

* Large amount of dark, coarse hair on the arms
* History of allergies to alpha hydroxy acids (AHAs), retinoids, soaps, fragrances, sunscreens or Latex
* Currently using over-the-counter AHA or retinol within one month or prescription retinoid within three months of the start of the study.
* History of skin cancer, including squamous or basal cell carcinoma at the treatment site or history of malignant melanoma.
* History of diabetes
* Currently pregnant or nursing

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Skin Collagen/Elastin ratio over time - Change from baseline in sun exposed, and non sun exposed skin areas. | up to 2 months
  The effects of tretinoin cream on human skin will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Balu, PhD, Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- Beckman Laser Institute Medical Clinic, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No